CLINICAL TRIAL: NCT05335772
Title: The Upper-limb Functional Rehabilitation in Chronic Stroke Patients: From Neuroimaging and Bio-humoral Biomarkers of a Personalized Action Observation Treatment Based on Virtual Reality to a Maximized and Predictable Rehabilitative Outcome.
Brief Title: VR-based Action Observation Treatment for Upper Limb Rehabilitation in Stroke: a Multimodal Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CNR Institute of Neuroscience, Parma (Other)
Collaborators: Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, Pietro Avanzini, P.I, Head of the Parma Research Unit of CNR Institute of Neuroscience, CNR Institute of Neuroscience, Parma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR-AOT-GR-2019
Record Dates: First submitted 2022-03-21; First posted 2022-04-19 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-AOT (Experimental): Experimental group, observing actions in virtual reality
  Interventions: Behavioral: Action Observation and following Action Execution
- VR-LO (Other): Control group, observing a matched dose of videos depicting landscapes in virtual reality
  Interventions: Behavioral: Landscape Observation and following Action Execution

INTERVENTIONS:
Behavioral: Action Observation and following Action Execution — VR-AOT patients will observe, rehearse and execute specific upper limb motor task belonging to activities of daily living.
  Arms: VR-AOT
Behavioral: Landscape Observation and following Action Execution — VR-LO participants will observe virtually explorable landscapes lasting for a matched duration. Then, they will be asked to actively perform the same set of hand actions requested to VR-AOT experimental groups.
  Arms: VR-LO

SUMMARY:
The loss of upper-limb motor functioning due to ischemic stroke has a negative impact on quality of life of patients. Action Observation Treatment (AOT), recently developed based on the mirror mechanism functioning, has proved effective in promoting plasticity into the motor system, ultimately boosting the motor recovery. The use of virtual reality further empowers the effectiveness of AOT, making the visual experience more first-person, and thus more realistic. A complete picture of the neurobiological mechanisms underlying AOT effectiveness is lacking to date, including the neuroradiological and biohumoral markers modulated by AOT, and their role in predicting the clinical outcome. Starting from these premises, the investigators propose a study aiming at evaluating the AOT effectiveness in post-stroke patients, and at identifying the biomarkers indexing the motor recovery process.

Sixty patients affected by ischemic stroke will be enrolled at Humanitas Clinical and Research Center IRCCS (ICH) Stroke Unit will be included and randomized in the following groups:

* VR-AOT: experimental group, observing actions in virtual reality
* VR-LO: control groups, observing a matched dose of videos depicting landscapes in virtual reality.

Clinical, neuroimaging and biohumoral evaluations, performed at Screening (Ts), Basal visit (T0), end-of-treatment (T1), 2 months follow up (FU-2), will include the following endpoints: Fugl-Meyer upper extremity motor scale (FM-UE); Nine-hole-peg test; Box and block test; Modified Ashworth scale; MRC; Pain Numeric-rating-scale; Functional Independence measure.

Patients will undergo treatment sessions for 6 weeks (5 days/week). VR-AOT patients will observe in virtual reality -rehearse and execute specific upper limb motor task belonging to activities of daily living. VR-LO participants will observe virtually explorable landscapes lasting for a matched duration. Then, participants will be asked to actively perform the same set of hand actions requested to VR-AOT experimental groups.

An intention-to-treat (ITT) analysis will be performed, using rmANOVA, minimal clinically important difference (MCID) in clinical outcomes, and chi-square test. For the primary endpoints, a two-arms rmANOVA with time as within-subject factor (3 levels: T0, T1, FU2) and group (VR-AOT vs VR-LO) as between-subjects factor will be conducted. The same approach will be adopted for secondary outcome measures. Subsequently, the effect of clinical, neuroradiological and biohumoral baseline features will be tested as regressors on the primary outcome variations via linear or ranked regression models. Significance will be set at 5%, and adjusted for MC.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Ischemic stroke in the territory of middle cerebral artery (MCA, lesion extension lower than half of its territory) or lacunar stroke
* MRC score 2-4 in at least one segment of the affected limb
* Modified Rankin Scale (mRS) prior to stroke ≤ 2
* Able to perform study requirements
* Able to give informed consent according to ICH/ GCP, and national/local regulations

Exclusion Criteria:

* Presence of global aphasia
* History of seizures
* Posterior circulation stroke
* Significant ipovisus
* Moderate-to severe neglect
* Cognitive impairment or language barriers
* Psychiatric comorbidities
* Drug or alcohol abuse
* Autoimmune disease
* Contraindication to perform MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Fugl-Meyer upper extremity motor scale at 6 weeks | Six weeks from baseline
  Stroke-specific, performance-based, impairment index (range 0-66, higher values indicate a better performance)

SECONDARY OUTCOMES:
Change from baseline Nine-hole-peg test at 6 weeks | Six weeks from baseline
  Standardized, quantitative test of upper extremity function
Change from baseline Nine-hole-peg test at 2 months | Two months from baseline
  Standardized, quantitative test of upper extremity function
Change from baseline Box and block test at 6 weeks | Six weeks from baseline
  Unilateral gross manual dexterity measure
Change from baseline Box and block test at 2 months | Two months from baseline
  Unilateral gross manual dexterity measure
Change from baseline Modified Ashworth Scale at 6 weeks | Six weeks from baseline
  Spasticity measure, evaluating limb's tone responsiveness to passive mobilization (Range: 0-4, higher values indicates higher degree of spasticity)
Change from baseline Modified Ashworth Scale at 2 months | Two months from baseline
  Spasticity measure, evaluating limb's tone responsiveness to passive mobilization (Range: 0-4, higher values indicates higher degree of spasticity)
Change from baseline Functional Independence Measure at 6 weeks | Six weeks from baseline
  Questionnaire measuring the independence in Activities of Daily Living (ADL). (Range: 18-126, higher values indicate an higher degree of functional independence)
Change from baseline Functional Independence Measure at 2 months | Two months from baseline
  Questionnaire measuring the independence in Activities of Daily Living (ADL). (Range: 18-126, higher values indicate an higher degree of functional independence)
Change from baseline Fugl-Meyer upper extremity motor scale at 2 months | Two months from baseline
  Stroke-specific, performance-based, impairment index (range 0-66, higher values indicate a better performance)

CONTACTS AND LOCATIONS:
Locations (1):
- Pietro Avanzini, Parma, Italy

IPD SHARING:
Plan to Share IPD: No